CLINICAL TRIAL: NCT03459664
Title: Evaluation of a Cross-sectional Coordinated, Severity Stepped, Evidence-based Care Model for Mental Disorders
Acronym: RECOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government); BARMER (Other); AOK Rheinland/Hamburg (Industry); DAK Gesundheit (Other); HEK (Unknown); BKK Linde (Unknown); BKK Mobil Oil (Industry); BKK Public (Unknown); BKK RWE (Unknown); BKK Salzgitter (Unknown); BKK Technoform (Unknown); BKK VerbundPlus (Unknown); Continentale BKK (Unknown); Heimat BKK (Unknown); Salus BKK (Unknown); TUI BKK (Unknown); WMF Betriebskrankenkasse (Unknown); IKK Classic (Unknown); Energie BKK (Unknown); VIACTIV Krankenkasse (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RECOVER
Record Dates: First submitted 2018-01-19; First posted 2018-03-09 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Delivery of Health Care
Keywords: stepped care; common mental disorders; managed care; integrated care; psychiatric disorders; psychotherapy; severe mental disorders
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with two arms (RECOVER or treatment as usual)
Who Masked: Outcomes Assessor
Masking Description: Individuals who evaluate the outcomes of interest will remain blinded regarding a participant's condition (RECOVER/TAU) over the course of the study. Randomization will be conducted after baseline assessment and communicated to the participant by a person that is not the outcome assessor. During follow-up assessments after 6 and 12 month the outcome assessor will remain blinded regarding a participant's condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RECOVER (Experimental): The intervention in the RECOVER stepped-care model includes specific evidence-based treatment options for severity grade 1 to 4.
  Interventions: Behavioral: RECOVER
- Treatment As Usual (Active Comparator): The active comparator is treatment as usual (TAU) and provides all common care options within the German health care system, depending on the severity grade 1 to 4.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: RECOVER — For each patient baseline assessment and individual support by a diagnostic and crisis resolution home treatment team is available. In addition, patients will be treated with specific interventions based on their severity grade:
  Grade 1 (mild): social support, information about mental disorder, e-therapy, consultation, self help, peer-support, supported employment.
  Grade 2 (medium): psychotherapy (stepped short-term and group therapy), if applicable medical treatment, e-therapy, peer-support, supported employment.
  Grade 3 (medium to severe): case management, psychotherapy (stepped short-term and group therapy), if applicable medical treatment, e-therapy, peer-support, supported employment.
  Grade 4 (severe): assertive community treatment, psychotherapy, medical treatment, e-therapy, peer-support, supported employment.
  Arms: RECOVER
Behavioral: Treatment as usual — For each patient all common care options within the German health care system are available, depending on the severity grade 1 to 4.
  This includes the following options: hospital based in-patient, out-patient treatment and day care, community based health care services, general practitioners, private psychiatrists and psychotherapists, self help.
  Arms: Treatment As Usual

SUMMARY:
This study evaluates a cross sectional, severity stepped, evidence-based care model for patients with mental disorders (RECOVER).

RECOVER is a consortium of well-known institutions for the treatment and integrated care of patients with mental disorders, patient associations, relative associations, research institutions, health care insurances and authorities from the care region Hamburg, Germany.

This project aims to evaluate the RECOVER care model with treatment as usual (TAU) regarding cost-effectiveness (costs, efficiency and cost utility) for patients with mental disorders.

The following questions are examined:

1. Does RECOVER reduce psychiatric health care costs compared to TAU?
2. Does RECOVER improve patient relevant outcomes (i.e. symptom remission, response, daily functioning and quality of life)?
3. Is RECOVER cost effective compared to TAU? (from a payer's and societal perspective)

A total sample of 890 patients with mental disorders will be assessed at baseline (before treatment) and randomized into the RECOVER care model or get TAU. Follow-up assessments are conducted after 6 month and 12 month.

As primary outcomes, cost reduction, improvement in symptoms (i.e. amount of remission and response to treatment, daily functioning and quality of life) and cost-efficiency-ratios will be measured. In addition, several secondary outcome parameters will be assessed.

Impact: The present randomized controlled trial (RCT) evaluates the cross-sectional, severity stepped, evidence-based approach of the RECOVER model in patients with mental disorders. With its focus on effectiveness and cost-effectiveness, the study aims to improve the health care system in Germany.

DETAILED DESCRIPTION:
Participants will be recruited from regular care settings (in-patient and out-patient services, general practitioners, psychotherapists) and via the RECOVER homepage. Upon fulfillment of the inclusion criteria and after having obtained informed consent, participants will undergo a complex baseline psychiatric diagnostic assessment, including among other measures the global assessment of functioning (GAF), severity of illness (CGI-S) and specification of diagnosis (SCID I and SCID II). Based on these three instruments, participants will be divided into four degrees severity: Grade 1 = mild, Grade 2 = medium, Grade 3 = medium to high, Grade 4 = severe mental disorder. Accordingly, there will be four strata of similar sample sizes (planned n=268, including 30% drop out rate; see power analysis below). Each participant will then be randomized either to the RECOVER treatment condition or the treatment as usual (TAU) condition. Randomization will be conducted by an independent person not involved in the RCT or diagnostic assessment, who will receive the pseudonymised participant ID and stratum number. A previously with the STATA 14 program defined list will be used to achieve randomization. When the planned sample size per stratum is achieved, no further patients will be included in this stratum.

For a complete list of measures, please refer to outcome measures section. In addition, secondary data will be obtained from external data owners, essential for the achievement of RECOVER's research objective - the determination of health costs. These include personal patient-related data such as data from health insurances companies (e.g. data from inpatient and outpatient medical services, rehabilitation services, transport, medical aid, drug/ medication data, home assistance and care services, work disability and sickness benefit/ allowance data). These will be inquired from the health insurance for the years 2016 to 2021 at the 12-month point in time and continuously assessed within the quality assurance study. Subsequently, a monetary valuation is carried out using standardized monetary valuation rates.

Serious adverse events (SAE) will be documented from the first contact (i.e. registry) between patient and study staff and will be included in the participant's record. A copy of each SAE protocol will be directly forwarded to the study's central management. Each SAE is assessed in terms of its causal relationship between the event and the study procedures (""serious undesirable, study-related event"). For each SAE, the SAE protocol must be filled in (with pseudonymised data only) and will be immediately discussed with the study management, who will check the protocol for plausibility and completeness and evaluate the event. Events that have not yet been formally completed are tracked. If the undesired event has been resolved, a final documentation is provided on the SAE protocol. The executive committee is informed by the study management and asked for an assessment. If all assessments have shown that the suspected case is an SAE, all study staff will be informed by the study management immediately, but at the latest within 7 days of notification.

The sample size is based on a power calculation to detect a statistically significant difference between the intervention (RECOVER) vs. standard care (TAU) in order to yield a small to medium standardized mean difference between the groups (Cohen's f of 0.175) after 12 months. At a power of at least 80% with a type 1 error rate of 5%, 2-sided testing and 10% of declared variance due to baseline, at least 233 study participants are required. For testing hypotheses involving the interaction of intervention and stratification subgroup, sample size increases to n=383. Diagnostics and therapy are carried out in approx. 50 clusters with approx. 21 participants each and an intraclass correlation (ICC) of .05 is assumed for the primary, continuous outcome. This results in a design effect of approximately 2.0 and a total sample size of 890 patients (including 30% dropout). With an estimated participation rate of 50%, 2140 patients must be addressed for participation.

Statistical analysis will be supervised by the local Department of Medical Biometry and Epidemiology. The analysis of primary and secondary outcome data is performed according to the intention-to-treat (ITT) principle. Missing values for the follow-up time points will be accounted for within mixed linear and logistic regression models. For sensitivity analyses, missing values will be replaced by multiple imputation and per-protocol (PP) analyses. The analysis of therapy utilization and productivity losses is performed descriptively as well as with difference-in-difference regressions (to analyze the measured costs over time). In addition, multivariate analyses will be carried out. Remission and response data are analyzed using logistic regression, while remission (non-clinical, i.e., performance under critical cut-off) and response (i.e. reduction in symptom severity of 50%) are specifically determined for each psychiatric condition during follow-up as compared to the baseline measurement. Changes in symptoms, level of functioning and health associated quality of life are analyzed with difference-in-difference-regression. To estimate cost efficiency, incremental cost-efficiency-relation (ICER) is calculated. To estimate the ICER's uncertainty, cost-efficiency-acceptance-curves based on net-benefit-regressions are calculated. All secondary outcome parameters are descriptively investigated as well as using multivariate analyses (e.g. logistic regression, difference-in-difference-regression). To assess inhibiting and promoting factors for the RECOVER model, qualitative measures are applied.

All study data are immediately entered into a database. To minimize input errors, all data are entered by two different staff members independently. During data entry, integrity checks are performed to minimize input errors. These tests are carried out on the basis of a data validation plan and are countersigned by the head of study and the study statistician. The data input system enables continuous quality control of the input process via integrated inspection functions.

After completion of the data entry, the access rights to the database are cancelled and the database is exported to the data transformation system. There, final plausibility checks are carried out and the data are checked for consistency and completeness. Missing values and inconsistencies are reported back to the examiner and processed by the person responsible. As soon as all corrections have been completed, the database is closed and transferred to the study statistician. All data entries, modifications or deletions are logged. All data (i.e. completed questionnaires, database) will be protected against unauthorized access, i.e. by physical locking in steel cabinets or secured by a system of individual access authorizations. In accordance with the principles of good clinical practice, all study data and relevant correspondence are archived by the investigators. Once the study has been completed, the all archived data will be stored by the University of Hamburg in accordance with legal regulations. The lead investigator is responsible for storing and archiving the study data.

Quality assurance will be achieved by evaluation and comparison of data assessed at baseline and at follow-up assessments after six month (t6) and after one year (t12). Data contains measures of disease symptoms and severity (e.g., HEALTH-49, CGI-S, PANSS, PHQ-9, GAD-7, PHQ-15, PID-5). The daily function level is measured with the GAF, and health-related quality of life is assessed with the EQ-5D-5L and the SF-12. Treatment satisfaction will also be measured. The therapeutic coherence is determined with regard to both drug and non-drug treatment. All therapeutic services will be continuously documented in terms of number, type and duration.

Data collection and monitoring will be carried out by treatment-unrelated, independent researchers (Dept. of Health Economics and Healthcare Research, Dept. of Medical Psychology and the Dept. of Medical Biometry and Epidemiology, UKE). They will primarily monitor compliance with the principles of good clinical practice and the study protocol, as well as proper data collection and input. Data verification will mainly focus on key variables that are defined at the beginning of the study. Frequency and duration of monitor visits will depend on recruitment progress, protocol compliance and data quality. It will be the monitor's responsibility to regularly check data collection and input, monitor adherence to the study protocol, and check that data are complete, consistent and correct. The monitor should have access to all data sources that can be used to verify the questionnaire information. In addition, in accordance with the regulations governing the monitoring of clinical trials, it is necessary for the investigator to grant the monitor access to the proportion of all pseudonymised patient files directly associated with the trial.

Study results as well as a detailed study protocol will be published in national and international peer-reviewed scientific journals. A publication agreement for the participating institutions will be achieved within a consortium agreement.

All data, personal identification data and scientific data, will be stored in the UKE's Dept. of Health Economics and Healthcare Research and Dept. of Medical Psychology for 10 years. Consent declarations will be stored in the study center's paper archive until a legally compliant scan is implemented. At all other locations, data will only be stored temporarily for immediate data processing as proposed within the study framework.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years
* insured in one of the relevant health insurances (BARMER GEK, AOK Rheinland/Hamburg, DAK Gesundheit, HEK, BKK Linde, BKK Mobil Oil, BKK Public, BKK RWE, BKK Salzgitter, BKK Technoform, BKK VerbundPlus, Continentale BKK, Heimat BKK, Salus BKK, TUI BKK, WMF Betriebskrankenkasse, IKK Classic, VIACTIV Krankenkasse)
* at least diagnosed with one of the relevant psychiatric disorders: Schizophrenic disorders (ICD-10: F20, F22, F23, F25); bipolar disorder (ICD-10: F31); major depressive disorder (ICD-10: F32, F33); anxiety disorder (ICD-10: F40, F41); obsessive compulsive disorder (ICD-10: F42); post traumatic stress disorder (ICD-10: F43.1); adjustment disorder (ICD-10: F43.2); somatoform disorder (ICD-10: F45); eating disorder (ICD-10: F50); personality disorder (ICD-10: F60, F61); attention-deficit hyperactivity disorders (ICD-10: F90);
* living in the surrounding area of the university medical center Hamburg-Eppendorf

Exclusion Criteria:

* disorder belonging to ICD-10 F0 (mental disorders due to known physiological conditions) or F1 (primary disorders due to psychoactive substance use)
* severe to most severe low intelligence (previously diagnosed ICD-10: F72/F73)
* insufficient language skills
* uncorrected visual and/or hearing impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
health care costs | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show a reduction in average health care costs. Different cost-sectors are assessed, with the Questionnaire for the Assessment of Medical and non-Medical Resource Utilisation in Mental Disorders (FIMPsy, Grupp et al., 2017) and the Questionnaire for the use of medical and non-medical services in old age (FIMA, Seidl et al., 2015), and will be added up to one measure "health care costs".
psycho-functional level | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an improvement in the psycho-functional level. The psycho-functional level is assessed as a combined outcome criterion (Aiken, 1987). For this purpose, scores of the Psychopathological Symptom Severity Scale of the Hamburg Modules for the Assessment of Psychosocial Health (HEALTH 49, Rabung, et al., 2007), the Global Assessment of Functioning Scale (GAF; Gold, 2014), and the Mental Component Summary of the Short Form Health-Questionnaire (SF-12, Ware et al., 1996) will be linearly transformed and added up to one measure "psycho-functional level".
incremental cost-effectiveness ratio (ICER) | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU shows an improvement in the incremental cost-effectiveness ratio (ICER). The ICER is calculated as the ratio of the difference in costs between RECOVER and TAU to the difference in quality adjusted-life years (QALYs) between RECOVER and TAU.

SECONDARY OUTCOMES:
severity of illness | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU lead to a greater reduction of severity of illness, assessed with the Clinical Global Impressions- Severity Scale (CGI-S; Guy 1976). The CGI-S requires a clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The following ratings are possible: 0 = not applicable; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill patients.
global functioning | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU lead to a greater improvement of global functioning, assessed with the Global Assessment of Functioning scale (GAF; Gold, 2014). GAF scores range from 100 (extremely high functioning) to 1 (severely impaired).
recovering quality of life | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU lead to a greater recovering quality of life, assessed with the Recovering Quality of Life questionnaire (Re-QOL-20, Keetharuth et al., 2017). Re-QOL-20 scores range from 0 to 80, where 0 indicates poorest quality of life and 80 indicates highest quality of life.
symptomatic remission | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show a higher proportion of symptomatic remission (number of patients). Symptomatic remission is defined according to Guy et al. (1975) with a value of ≤ 3 points in the severity score of clinical global impression scale (no greater than "mild") for ≥ 6 months.
functional remission | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show a higher proportion of functional remission (number of patients). Functional remission according to the criterion by Albert et al. (2012), measured with the global assessment of functioning scale (GAF; Gold, 2014) fulfilled when a value of ≥ 60 points persisted for ≥ 6 months.
rate of psychiatric hospitalizations | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show a reduction of psychiatric hospitalizations (number of hospitalizations since baseline)
duration of psychiatric hospitalizations | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show a reduction in the duration of psychiatric hospitalizations (number of days in hospitalizations since baseline)
incapacity to work | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show a reduction in incapacity to work (number of days since baseline)
delay of treatment | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show a reduction in delay of diagnosis specific treatment (number of days between baseline and start of treatment).
evidence-based interventions | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an increase of guideline directed treatment, according to specific diagnosis and severity grade (number of patients with guideline directed treatment)
out-patient psychotherapeutic interventions for severe mental disorders | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an increase of patients with severe mental disorders in out-patient psychotherapeutic interventions (number of patients)
psychotherapeutic group interventions | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an increase of group psychotherapeutic interventions (number of patients)
psychotherapeutic short-term interventions | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an increase of psychotherapeutic short-tern interventions (number of patients)
specific psychiatric interventions for severe mental disorders | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an increase of specific psychiatric interventions for severe mental disorders (number of crisis resolution and assertive community treatment)
treatment retention | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an improvement in treatment retention rate (days until drop out after baseline)
drop out rate | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an improvement in drop-outs during treatment (number of drop outs)
web-based therapy | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an improvement in utilization of web-based therapy (number of users).
peer-support | Baseline, 12 month after baseline
  Inclusion in the treatment arm of the RECOVER trial for a maximum of 12 month from baseline compared to TAU show an improvement in utilization of peer-support (number of users)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Peth, Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Institute and Outpatients Clinic Medical Psychology; Holger Schulz, Prof., Principal Investigator — University Medical Center Hamburg-Eppendorf, Institute and Outpatients Clinic Medical Psychology; Hans-Helmut König, Prof., Principal Investigator — Institute of Health Economics and Health Care Research
Locations (1):
- University Medical Center Hamburg-eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schindler A, Warkentin HF, Bierbrodt J, Konig H, Konnopka A, Pepic A, Peth J, Lambert M, Gallinat J, Karow A, Konig HH, Harter M, Schulz H, Rohenkohl A, Krog K, Biedermann SV, Schafer I. Dialectical behavior therapy (DBT) in an assertive community treatment structure (ACT): testing integrated care borderline (ICB) in a randomized controlled trial (RECOVER). Borderline Personal Disord Emot Dysregul. 2024 Aug 14;11(1):18. doi: 10.1186/s40479-024-00261-4. PMID 39138537
- [Derived] Konig H, Konig HH, Gallinat J, Lambert M, Karow A, Peth J, Schulz H, Konnopka A. Excess costs of mental disorders by level of severity. Soc Psychiatry Psychiatr Epidemiol. 2023 Jun;58(6):973-985. doi: 10.1007/s00127-022-02298-8. Epub 2022 May 31. PMID 35639134
- [Derived] Lambert M, Karow A, Gallinat J, Ludecke D, Kraft V, Rohenkohl A, Schroter R, Finter C, Siem AK, Tlach L, Werkle N, Bargel S, Ohm G, Hoff M, Peter H, Scherer M, Mews C, Pruskil S, Luke J, Harter M, Dirmaier J, Schulte-Markwort M, Lowe B, Briken P, Peper H, Schweiger M, Mosko M, Bock T, Wittzack M, Meyer HJ, Deister A, Michels R, Herr S, Konnopka A, Konig H, Wegscheider K, Daubmann A, Zapf A, Peth J, Konig HH, Schulz H. Study protocol for a randomised controlled trial evaluating an evidence-based, stepped and coordinated care service model for mental disorders (RECOVER). BMJ Open. 2020 May 4;10(5):e036021. doi: 10.1136/bmjopen-2019-036021. PMID 32371520
- See also: Homepage of the RECOVER model — https://www.recover-hamburg.de/